CLINICAL TRIAL: NCT04844450
Title: A Double-Blind, Placebo-Controlled, Randomized, Multipart, Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneously Administered JNJ-75220795
Brief Title: A Single and Multiple Ascending Dose Study of Subcutaneously Administered JNJ-75220795
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CR108997; 75220795NAS1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-04-13; First posted 2021-04-14 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose (SAD) (Experimental): Participants in cohorts 1-5 and cohorts 3a-5a will receive subcutaneous (SC) injection of single dose (Part A) of JNJ-75220795 or matching placebo.
  Interventions: Drug: JNJ-75220795; Drug: Placebo
- Multiple Ascending Dose (MAD) (Experimental): Participants in cohorts 6-8 will receive SC injection of 2 doses (Part B) of JNJ-75220795 or matching placebo. Participants in cohorts 9-11 will receive SC injection of 4 doses (Part C) of JNJ-75220795 or matching placebo.
  Interventions: Drug: JNJ-75220795; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-75220795 — JNJ-75220795 will be administered subcutaneously.
Drug: Placebo — Matching placebo will be administered subcutaneously.

SUMMARY:
The purpose of the study is to assess the safety and tolerability of single and multiple subcutaneous (SC) doses of JNJ-75220795.

ELIGIBILITY:
Inclusion Criteria:

* Participants with certain genetic predisposition to non-alcoholic fatty liver disease (NAFLD) determined at screening
* Presence of liver steatosis at screening
* Participants on anti-hypertensive and/or lipid lowering medications and/or glucose lowering medications must be on stable dose(s) for at least 4 weeks prior to screening
* Weight stable defined as no more than 5% body weight loss or gain within 3 months prior to screening and no more than 5% body weight loss or gain from screening to randomization

Exclusion Criteria:

* Known allergies, hypersensitivity, or intolerance to JNJ-75220795 or its excipients
* History of hepatitis B surface antigen (HbsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HbsAg or anti-HCV at screening
* History of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV at screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Signs and Symptoms/ Adverse Events (AEs) | Up to Day 182
  Number of participants with treatment-emergent signs and symptoms/adverse events (including allergic reactions/hypersensitivity and local injection site reactions) will be reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Treatment-emergent adverse events (TEAEs) are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Number of Participants With Change From Baseline in Vital Signs Abnormalities | Baseline, up to Day 168
  Number of participants with change from baseline in vital signs abnormalities including temperature, heart rate, respiratory rate, and blood pressure (supine) will be reported.
Number of Participants With Change From Baseline in Clinical Laboratory Abnormalities | Baseline, up to Day 168
  Number of participants with change from baseline in clinical laboratory abnormalities including hematology, chemistry and urinalysis will be reported.
Number of Participants With Change From Baseline in Physical Examination Abnormalities | Baseline, up to Day 168
  Number of participants with change from baseline in physical examination abnormalities will be reported.
Number of Participants With Change From Baseline in Electrocardiogram (ECG) Abnormalities | Baseline, up to Day 168
  Number of participants with change from baseline in ECG abnormalities will be reported.

SECONDARY OUTCOMES:
Percent Change From Baseline in Liver Fat Content | Baseline, weeks 6, 12, 18 and 24
  Percent change from baseline in liver fat content will be reported.
Plasma Concentration of JNJ-75220795 Over Time | SAD: Predose, up to Day 3 and MAD: Predose, up to Day 86
  Plasma samples will be analyzed to determine concentrations of JNJ-75220795.
Percentage of Participants With Treatment-emergent Anti Drug Antibodies (ADA) | Up to Day 168
  Percentage of participants with treatment-emergent ADA will be assessed using a validated assay for ADA analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- United States (2):
  - Research Centers of America, LLC, Hollywood, Florida
  - Endeavor Clinical Trials, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Wang C, Guo P, Liu X, Xu X, Zou L, Meng S, Guo Q, Wen Q, Yang C. Association Between PNPLA3 Inhibition and Gout: A Drug Target Mendelian Randomization Study. Int J Endocrinol. 2025 Aug 20;2025:6664846. doi: 10.1155/ije/6664846. eCollection 2025. PMID 40881642